CLINICAL TRIAL: NCT00518960
Title: The Effects of ProAlgaZyme Novel Algae Infusion on HDL Cholesterol and C-Reactive Protein in Individuals With Metabolic Syndrome
Brief Title: The Effects of ProAlgaZyme on HDL Cholesterol in Individuals With Metabolic Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Health Enhancement Products, Inc. (Industry)
Collaborators: MAPS Applied Research Center (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-0003-02; MARC007-003
Record Dates: First submitted 2007-08-17; First posted 2007-08-21 (Estimated); Last update posted 2007-08-21 (Estimated); Status verified 2007-08

CONDITIONS: Metabolic Syndrome; Hyperlipidemia
Keywords: ProAlgaZyme; Algae; High density lipoprotein; HDL; C-Reactive Protein; CRP; Hyperlipidemia; Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome; Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ProAlgaZyme

SUMMARY:
The purpose of this study is to determine the effectiveness of ProAlgaZyme in increasing levels of HDL 'good' cholesterol and decreasing total cholesterol and C-reactive protein in patients with Metabolic Syndrome.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the most common cause of mortality in the United States. In 1988, Reaven, et al. published findings that indicate a majority of individuals who developed CVD had multiple concurrent risk factors including dyslipidemia, hypertension, and hyperglycemia. Reaven, et al., defined this cluster of risk factors as Syndrome X and hypothesized that insulin resistance was the underlying factor in its development. Over time, metabolic syndrome has been used as a more meaningful term and additional risk factors have been associated with its diagnosis (Grundy, et al. 2004). Metabolic syndrome is an increasingly prevalent problem in the United States and other westernized nations. It is estimated that approximately 50 million Americans have metabolic syndrome. The risk factors linked to metabolic syndrome include:

* Abdominal obesity
* Atherogenic dyslipidemia (high triglycerides, low HDL cholesterol and high LDL cholesterol)
* Elevated blood pressure
* Insulin resistance with or without glucose intolerance
* Pro-thrombotic state (e.g., high fibrinogen or plasminogen activator inhibitor-1 in the blood)
* Pro-inflammatory state [e.g. elevated C-reactive protein (CRP)in the blood]

The management goals for metabolic syndrome include reducing the risk for developing CVD and type 2 diabetes. Therefore, therapy is directed at reducing LDL cholesterol, blood pressure and glucose as well as increasing HDL cholesterol levels. Additional interventions to control blood pressure and lipids provide the next line of treatment for patients with metabolic syndrome.

ProAlgaZyme, a novel fermentation product of a freshwater algae ecosystem, will be evaluated in this trial for its effects on circulating lipids. According to the sponsor, ProAlgaZyme is expected to increase the circulating levels of HDL cholesterol while lowering total cholesterol and CRP. ProAlgaZyme was previously tested in a double blind, placebo controlled, pilot trial in 60 subjects with metabolic syndrome (30 subjects per arm), conducted at the University of Yaoundé, Cameroon. Statistically significant (p < 0.05 or better) improvements were seen in total cholesterol, HDL-C and C-reactive protein when compared to placebo. (In Press - Lipids in Health and Disease)

The present study will evaluate the effect of ProAlgaZyme versus placebo on blood lipids and hsCRP in subjects who meet the criteria for Metabolic Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 28-40
* Subjects with at least 3 of the following parameters:

  * Elevated waist circumference: Men - Equal to or greater than 40 in (102cm); Women - Equal to or greater than 35 in (88cm)
  * Elevated triglycerides: Equal to or greater than 150 mg/dL
  * Reduced HDL ("good") cholesterol: Men - Less than 40 mg/dL; Women - Less than 50 mg/dL
  * Elevated blood pressure: Equal to or greater than 130/85 mmHg
  * Elevated fasting glucose: Equal to or greater than 100 mg/dL
  * Elevated CRP: Equal to or greater than 5 mg/L
* Subjects with ability to comprehend and complete the questionnaires and forms
* Subjects whose schedules permit 4 visits to the study center over the duration of the trial
* Subjects who are likely to comply with study procedures and test article consumption
* Subjects who are likely to abstain from taking unauthorized supplements/medications or participating in any other clinical trial or experimental treatment during this trial

Exclusion Criteria:

* Subjects with uncontrolled hypertension as defined as greater than 180/95 mmHg (subjects may be re-screened after adequate blood pressure control has been maintained)
* Women who are pregnant or lactating, or who are of child-bearing potential and not using an acceptable method of birth control
* Subjects with a history of hepatic or renal disease, insulin dependent diabetes, active cancer, HIV infection or blood dyscrasias
* Current use of lipid-lowering medications, anti-inflammatories such as low-dose aspirin, or herbal therapies known to affect inflammation or blood lipids 8 weeks prior to study entry
* Current use of Metformin
* More than moderate alcohol use (> 14 drinks per week)
* Use of illicit drugs
* Acute coronary syndrome, heart failure, CVA, or coronary intervention within 6 months prior to study
* Serious or unstable medical or psychological conditions that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-04; Study Completion 2007-09 (Estimated)

PRIMARY OUTCOMES:
HDL Cholesterol | 12 weeks

SECONDARY OUTCOMES:
Lipid Panel (Total Chol., LDL-Chol., Triglycerides, Total Chol./HDL-Chol. ratio) | 12 weeks
C-Reactive Protein | 12 weeks
Blood Pressure | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Terence Pertile, Ph.D., Principal Investigator — MAPS Applied Research Center
Locations (1):
- MAPS Applied Research Center (MARC), Edina, Minnesota, United States